CLINICAL TRIAL: NCT03255733
Title: Intense Therapeutic Ultrasound for Chronic, Subcutaneous Lateral Epicondylitis Musculoskeletal Pain Reduction
Brief Title: ITU Treatment for Chronic Epicondylitis Musculoskeletal Pain Reduction
Acronym: ITU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guided Therapy Systems (Industry)
Collaborators: More Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GTS-ITU Epicondylosis 01
Record Dates: First submitted 2017-08-10; First posted 2017-08-21 (Actual); Results first posted 2017-11-17 (Actual); Last update posted 2017-11-17 (Actual); Status verified 2017-10

CONDITIONS: Tennis Elbow
Keywords: Chronic Lateral Epicondylitis; Tennis Elbow; Intense Therapeutic Ultrasound (ITU); Guided Therapy Systems (GTS); Ardent Sound, Inc.; Actisound
MeSH Terms: conditions — Tennis Elbow

STUDY DESIGN:
Intervention Model Description: Patients age 18 - 85, previously diagnosed with Chronic Lateral Epicondylitis, with symptoms exceeding 90 days, and where Standard of Care treatments have failed to resolve the symptoms.
Masking Description: Investigator was blinded to the Patient Reported Outcome Measure Survey details and analysis.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Intense Therapeutic Ultrasound Treatment (Experimental): Intense Therapeutic Ultrasound applied along and length and width of the Common Extensor Tendon. 80, 1 Joule pulses were applied twice, four weeks apart.
  Interventions: Device: Intense Therapeutic Ultrasound Treatment

INTERVENTIONS:
Device: Intense Therapeutic Ultrasound Treatment
  Other Names: Guided Therapy Systems, Ardent Sound, GTS, ITU; Actisound

SUMMARY:
This study evaluates the effectiveness, safety and patient tolerance for the use of Intense Therapeutic Ultrasound (ITU) for chronic, subcutaneous lateral Epicondylitis musculoskeletal tissue pain reduction began in July 2015 and was completed in March 2017. The More Foundation/The Core Institute: Single-blinded pivotal study for the treatment of chronic lateral epicondylitis. A total 29 patients received 2 treatments, 4 weeks apart on subcutaneous musculoskeletal tissues along with Standard of Care treatments as prescribed by the Principal Investigator. Patients were followed for up to 6 months after the first treatment receiving a physical exam at each follow-up visit (4, 8 and 12 weeks) and provided feedback via Patient/Subject Reported Outcome Measure surveys specific to the treated anatomy at each visit and via phone follow-up at 26 weeks after the first treatment.

DETAILED DESCRIPTION:
Intense therapeutic ultrasound (ITU) is an established ultrasound based therapy in which sound waves are concentrated and focused into selected musculoskeletal tissue, to produce selective thermal coagulative changes over a small controlled area while leaving the surrounding tissue unaffected. These coagulative changes are known to begin the body's tissue response cascade and promote collagen generation in the targeted anatomy resulting in pain reduction.

ITU has been used clinically for treating the subcutaneous musculoskeletal tissue below facial skin for the past decade and it has received CE Mark and FDA 510(k) clearance to market for non-surgical brow and submental tissue lifting. Over 3 Million patients worldwide have been treated using this technology. Clinical studies have shown that 85% of patients receiving this treatment on facial skin tissue showed an improvement in facial lifting with no significant pain, erythema, inflammation or scarring by creating the same coagulative changes to the connective tissue under the skin. Histologically, it has been shown that ITU induces the production of dermal collagen with thickening of the dermis and straightening of the elastic fibers in the reticular dermis.

On-going research in laboratory studies has shown that ITU can improve healing of damaged Achilles tendon in a rabbit model. Preliminary results showed an increase in precursor markers for collagen regeneration (e.g. Vascular endothelial growth factor A (VEGFa), tumor necrosis factor alpha (TNFα), Interleukin 1 beta (IL-1β), and Transforming growth factor beta 1 (TGFβ1)) and subsequent increase in collagen formation in injured rabbit tendons treated with ITU compared to injured, untreated rabbit tendons.

ELIGIBILITY:
Inclusion Criteria:

* Chronic Pain (>90 days) from previously diagnosed Lateral Epicondylitis, where "Standard of Care" regimens failed to relief pain in the affected anatomy.
* No History of surgery to the affected anatomy.
* No alternative treatment procedures within the last 90 days.
* Unilateral Pain
* Willingness to complete treatment and post treatment regimen as described.
* Patients who have provided written and verbal informed consent.

Exclusion Criteria:

* Patients currently enrolled in any other non-conservative, device, or Investigational New Device (IND) clinical trial, or who have participated in a clinical study involving the Common Extensor Tendon, thirty days prior to study initiation;
* Patients who have participated in any other clinical study involving an investigational product 30 days prior to enrollment that, in the opinion of the Principal Investigator, could affect the outcome of this study;
* Patients who have received previous treatment in the symptomatic limb (not including conservative treatment);
* At the Principal Investigator's discretion, any patient that should be excluded based on their current condition or medical history.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2015-07-14 (Actual); Primary Completion 2017-03-13 (Actual); Study Completion 2017-03-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John A Kearney, MD, Principal Investigator — The More Foundataion
Locations (1):
- The More Foundation, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] White WM, Makin IR, Barthe PG, Slayton MH, Gliklich RE. Selective creation of thermal injury zones in the superficial musculoaponeurotic system using intense ultrasound therapy: a new target for noninvasive facial rejuvenation. Arch Facial Plast Surg. 2007 Jan-Feb;9(1):22-9. doi: 10.1001/archfaci.9.1.22. PMID 17224484
- [Background] Alam M, White LE, Martin N, Witherspoon J, Yoo S, West DP. Ultrasound tightening of facial and neck skin: a rater-blinded prospective cohort study. J Am Acad Dermatol. 2010 Feb;62(2):262-9. doi: 10.1016/j.jaad.2009.06.039. PMID 20115948
- [Background] Gliklich RE, White WM, Slayton MH, Barthe PG, Makin IR. Clinical pilot study of intense ultrasound therapy to deep dermal facial skin and subcutaneous tissues. Arch Facial Plast Surg. 2007 Mar-Apr;9(2):88-95. doi: 10.1001/archfaci.9.2.88. PMID 17372061
- [Background] Laubach HJ, Makin IR, Barthe PG, Slayton MH, Manstein D. Intense focused ultrasound: evaluation of a new treatment modality for precise microcoagulation within the skin. Dermatol Surg. 2008 May;34(5):727-34. doi: 10.1111/j.1524-4725.2008.34196.x. PMID 18429926
- [Background] Molloy T, Wang Y, Murrell G. The roles of growth factors in tendon and ligament healing. Sports Med. 2003;33(5):381-94. doi: 10.2165/00007256-200333050-00004. PMID 12696985
- [Background] Charan J, Biswas T. How to calculate sample size for different study designs in medical research? Indian J Psychol Med. 2013 Apr;35(2):121-6. doi: 10.4103/0253-7176.116232. PMID 24049221
- [Background] DiGiovanni BF, Nawoczenski DA, Lintal ME, Moore EA, Murray JC, Wilding GE, Baumhauer JF. Tissue-specific plantar fascia-stretching exercise enhances outcomes in patients with chronic heel pain. A prospective, randomized study. J Bone Joint Surg Am. 2003 Jul;85(7):1270-7. doi: 10.2106/00004623-200307000-00013. PMID 12851352
- [Background] Rompe JD, Overend TJ, MacDermid JC. Validation of the Patient-rated Tennis Elbow Evaluation Questionnaire. J Hand Ther. 2007 Jan-Mar;20(1):3-10; quiz 11. doi: 10.1197/j.jht.2006.10.003. PMID 17254903

RESULTS

PARTICIPANT FLOW:
Groups:
- Intense Therapeutic Ultrasound Treatment: Intense Therapeutic Ultrasound applied along and length and width of the Common Extensor Tendon. 80, 1 Joule pulses were applied twice, four weeks apart.
  Intense Therapeutic Ultrasound Treatment
Period: Overall Study
Arm/Group | Intense Therapeutic Ultrasound Treatment
Started | 29
Completed | 25
Not Completed | 4
Not completed — Lost to Follow-up | 4

BASELINE CHARACTERISTICS:
Arm/Group | Intense Therapeutic Ultrasound Treatment
Number analyzed (Participants) | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 28
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 17
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 29

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Reporting at Least 25% Overall Pain Reduction
Description: Percentage of Patients Reporting at least 25% pain reduction compared to baseline, using Universal Visual Analog Scale (VAS) Pain Score. VAS is a 10-point Pain Scale, where 0 = No Pain, 1 = Slight Pain and 10 = the Patients Worst Imaginable Pain. Scales in between represent 10% increments of Pain ( Range 1 - 10).
Time Frame: 12 weeks after 1st Treatment
Population: Percentage of Patients reporting at least 25% improvement in Pain at 12 Weeks after the first treatment
Measure: Number; unit: percentage of patients with less pain
Arm/Group | Intense Therapeutic Ultrasound Treatment
Number analyzed (Participants) | 25
percentage of patients with less pain | 88

2. Secondary Outcome: Average Pain Score Change as Reported Using Patient Rated Tennis Elbow Evaluation, During Normal Activities
Description: Average Percentage of Pain Change as Reported using Patient-Rated Tennis Elbow Evaluation Survey, compared to baseline. Range (± 100%)
Time Frame: 12 weeks after 1st Treatment
Measure: Mean (Full Range); unit: percentage of reported pain change
Arm/Group | Intense Therapeutic Ultrasound Treatment
Number analyzed (Participants) | 25
percentage of reported pain change | -58 [-100 to 100]

ADVERSE EVENTS:
Time Frame: 2 Years
Description: Any self-reported adverse event occurring after the first treatment
Arm/Group | Intense Therapeutic Ultrasound Treatment
All-Cause Mortality (participants affected / at risk) | 0/29
Serious Adverse Events (participants affected / at risk) | 0/29
Other Adverse Events (participants affected / at risk) | 0/29

LIMITATIONS AND CAVEATS:
While the protocol involved Chronic patients, who had already failed Standard of Care regimens, it is a limitation for this investigational study to have no control group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2015-05-04): https://cdn.clinicaltrials.gov/large-docs/33/NCT03255733/Prot_000.pdf
  • Statistical Analysis Plan (2015-03-02): https://cdn.clinicaltrials.gov/large-docs/33/NCT03255733/SAP_001.pdf
  • Informed Consent Form (2015-03-02): https://cdn.clinicaltrials.gov/large-docs/33/NCT03255733/ICF_002.pdf